CLINICAL TRIAL: NCT00206076
Title: CellCept (Mycophenolate Mofetil, MMF) Maintenance Immunosuppression in Liver Transplant Recipients With Long-term Follow-up Post-transplantation for Non-Autoimmune Liver Disease - A Prospective, Randomized, Multicenter Trial.
Brief Title: Mycophenolate Mofetil Immunosuppression Without/With Reduced Dose Calcineurin Inhibitor Long After Liver Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEL350
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-07

CONDITIONS: Liver Disease
Keywords: Liver transplantation; Calcineurin inhibitor withdraw; mycophenolate mofetil; Immunosuppression side effects; Graft rejection
MeSH Terms: conditions — Liver Diseases | interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): mycophenolate mofetil monotherapy
  Interventions: Drug: mycophenolate mofetil
- 2 (Active Comparator): mycophenolate mofetil and half their baseline dose of calcineurin inhibitor
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: mycophenolate mofetil — mycophenolate mofetil and half their baseline dose of calcineurin inhibitor
  Arms: 2
Drug: mycophenolate mofetil — mycophenolate mofetil monotherapy
  Arms: 1

SUMMARY:
The purpose of the study is to assess the safety and efficacy of mycophenolate mofetil alone, or with reduced dose cyclosporine (CsA) or tacrolimus, for immunosuppression long-term after liver transplantation, in an attempt to reduce the potential side effects from using cyclosporine or tacrolimus.

DETAILED DESCRIPTION:
Most liver transplant recipients receive an immunosuppressive drug regimen that contains either cyclosporine or tacrolimus. Although these drugs have revolutionized transplantation, in many patients their long-term use is a major cause of serious side effects, including kidney failure, hypertension, diabetes mellitus, hyperlipidemia, and/or neurologic side effects. Stopping or reducing the dose of cyclosporine or tacrolimus can ameliorate the above side effects but may increase the risk of rejection. Mycophenolate mofetil (MMF), a safe and effective immunosuppressant that does not cause the above side effects, is typically used in combination with cyclosporine or tacrolimus. Attempts in liver transplant recipients at using mycophenolate mofetil alone or with reduced dose cyclosporine or tacrolimus have been successful but some patients developed rejection, and a few patients suffered liver failure. Most rejections after liver transplantation are easy to successfully treat with increased immunosuppression, but such treatment may carry risks such as increased susceptibility to infection. There have not yet been any large trials to adequately assess the safety and efficacy of using mycophenolate mofetil this way (alone or with reduced dose calcineurin inhibitor (CNI)).

The purpose of this trial is to evaluate whether mycophenolate mofetil as monotherapy or with reduced dose cyclosporine or tacrolimus long-term after liver transplantation is safe and decreases side effects related to calcineurin inhibitor use.

Only liver recipients expected to have a relatively low risk of developing rejection and/or liver failure are eligible for this trial. Some reasons for considering them low risk are their stable liver function, having had the transplant for over a year, having had one or fewer prior rejection episodes, having had non-autoimmune liver disease, their currently requiring low dose/level cyclosporine or tacrolimus, and the plan to use high dose mycophenolate mofetil and to exclude patients that fail to attain target values for mycophenolic acid area under the concentration-time curve (MPA AUC - MycoPhenolic Acid Area Under the Curve).

Eligible patients will be randomized to receive either mycophenolate mofetil monotherapy (MMF; CNI discontinued), or mycophenolate mofetil and half their baseline dose of calcineurin inhibitor (MMF; CNI decreased). The primary outcome is biopsy proven rejection and the secondary outcomes include patient and graft survival, adverse events, hepatic profile, blood pressure, renal function, diabetes, and lipid profile. Additionally, mycophenolic acid concentrations will be measured; a mycophenolate mofetil monotherapy trial provides unique opportunity to study the implications of such monitoring. Patients will be followed for 12 months; there will be 16 visits during the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age or older (females who can become pregnant must use two acceptable methods of birth control while taking mycophenolate mofetil)
* Orthotopic liver transplant more than one year prior to enrollment
* Using calcineurin inhibitor to prevent rejection at time of screening
* Patients must be willing to provide informed consent and abide by the requirements of the study

Exclusion Criteria:

* Liver disease may not have been secondary to an autoimmune cause, including:

  * autoimmune hepatitis,
  * primary sclerosing cholangitis,
  * primary biliary cirrhosis
* Patients who have had:

  * more than one prior episode of rejection,
  * rejection within the past six months,
  * any corticosteroid resistant rejection
* Patients with a tacrolimus trough level of greater than 7 ng/ml within 90 days prior to enrollment
* Patients with a cyclosporine trough level greater than 225 ng/ml within 90 days prior to enrollment
* Patients taking more the 5 mg per day of prednisone within 90 days prior to enrollment
* Patients taking any prednisone within 30 days of enrollment
* Allograft dysfunction within 6 months of enrollment, including ALT and/or total bilirubin greater than 2x normal, and/or biopsy proven hepatitis C virus (HCV) with fibrosis greater than stage II
* White blood cell count less than 2,500 or platelet count less than 50,000 within 60 days of enrollment
* MPA AUC threshold: Patients are not eligible for the study if they do not attain the threshold value MPA AUC (>30 mg*h/L if on CsA, >40 mg*h/L if on tacrolimus) after 50% calcineurin inhibitor reduction, measured using a 3-sample estimate (trough, 30-min, 120-min)
* Patients who have had a previous transplant of organ(s) other than liver
* Patients who received a liver from a hepatitis C positive donor
* Patients who received a liver from a living donor
* Patients with any technical complication requiring intervention within the three months prior to screening
* Current infection requiring treatment
* History of post transplant lymphoproliferative disorder
* History of malignancy other than non-melanoma skin cancer or Stage 1-2 hepatoma
* Active or unhealed duodenal ulcer
* Concomitant treatment with rapamycin and/or interferon
* Known allergy or sensitivity to CellCept® or any of its components
* Unable or unwilling to comply with the protocol requirements or considered by the investigator(s) to be unfit for the study
* Participation in a clinical trial within 30 days prior to study entry or prior enrollment in any CellCept® clinical trial
* Pregnant or breastfeeding woman
* Diabetes with known, clinically significant gastroparesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-08; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Reich, MD, Principal Investigator — Drexel College of Medicine
Locations (3):
- United States (3):
  - University of Kentucky at Lexington, Lexington, Kentucky
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Texas Transplant Institute, San Antonio, Texas

REFERENCES:
- [Background] Reich DJ, Clavien PA, Hodge EE; MMF Renal Dysfunction after Liver Transplantation Working Group. Mycophenolate mofetil for renal dysfunction in liver transplant recipients on cyclosporine or tacrolimus: randomized, prospective, multicenter pilot study results. Transplantation. 2005 Jul 15;80(1):18-25. doi: 10.1097/01.tp.0000165118.00988.d7. PMID 16003228
- [Background] Reich D, Rothstein K, Manzarbeitia C, Munoz S. Common medical diseases after liver transplantation. Semin Gastrointest Dis. 1998 Jul;9(3):110-25. PMID 9700842
- [Background] Mazariegos GV, Reyes J, Marino IR, Demetris AJ, Flynn B, Irish W, McMichael J, Fung JJ, Starzl TE. Weaning of immunosuppression in liver transplant recipients. Transplantation. 1997 Jan 27;63(2):243-9. doi: 10.1097/00007890-199701270-00012. PMID 9020325
- [Background] McDiarmid SV, Farmer DA, Goldstein LI, Martin P, Vargas J, Tipton JR, Simmons F, Busuttil RW. A randomized prospective trial of steroid withdrawal after liver transplantation. Transplantation. 1995 Dec 27;60(12):1443-50. doi: 10.1097/00007890-199560120-00013. PMID 8545872
- [Background] Fraser GM, Grammoustianos K, Reddy J, Rolles K, Davidson B, Burroughs AK. Long-term immunosuppression without corticosteroids after orthotopic liver transplantation: a positive therapeutic aim. Liver Transpl Surg. 1996 Nov;2(6):411-7. doi: 10.1002/lt.500020602. PMID 9346686
- [Background] Stegall MD, Everson GT, Schroter G, Karrer F, Bilir B, Sternberg T, Shrestha R, Wachs M, Kam I. Prednisone withdrawal late after adult liver transplantation reduces diabetes, hypertension, and hypercholesterolemia without causing graft loss. Hepatology. 1997 Jan;25(1):173-7. doi: 10.1002/hep.510250132. PMID 8985286
- [Background] Hodge EE, Reich DJ, Clavien PA, Kim-Schluger L. Use of mycophenolate mofetil in liver transplant recipients experiencing renal dysfunction on cyclosporine or tacrolimus-randomized, prospective, multicenter study results. Transplant Proc. 2002 Aug;34(5):1546-7. doi: 10.1016/s0041-1345(02)03014-2. No abstract available. PMID 12176477
- [Background] Raimondo ML, Dagher L, Papatheodoridis GV, Rolando N, Patch DW, Davidson BR, Rolles K, Burroughs AK. Long-term mycophenolate mofetil monotherapy in combination with calcineurin inhibitors for chronic renal dysfunction after liver transplantation. Transplantation. 2003 Jan 27;75(2):186-90. doi: 10.1097/01.TP.0000041702.31262.CD. PMID 12548120
- [Background] Schlitt HJ, Barkmann A, Boker KH, Schmidt HH, Emmanouilidis N, Rosenau J, Bahr MJ, Tusch G, Manns MP, Nashan B, Klempnauer J. Replacement of calcineurin inhibitors with mycophenolate mofetil in liver-transplant patients with renal dysfunction: a randomised controlled study. Lancet. 2001 Feb 24;357(9256):587-91. doi: 10.1016/s0140-6736(00)04055-1. PMID 11558484
- [Background] Herrero JI, Quiroga J, Sangro B, Girala M, Gomez-Manero N, Pardo F, Alvarez-Cienfuegos J, Prieto J. Conversion of liver transplant recipients on cyclosporine with renal impairment to mycophenolate mofetil. Liver Transpl Surg. 1999 Sep;5(5):414-20. doi: 10.1002/lt.500050513. PMID 10477843
- [Background] Stewart SF, Hudson M, Talbot D, Manas D, Day CP. Mycophenolate mofetil monotherapy in liver transplantation. Lancet. 2001 Feb 24;357(9256):609-10. doi: 10.1016/s0140-6736(00)04065-4. PMID 11558493
- [Background] Munoz SJ, Rothstein KD, Reich D, Manzarbeitia C. Long-term care of the liver transplant recipient. Clin Liver Dis. 2000 Aug;4(3):691-710. doi: 10.1016/s1089-3261(05)70133-1. PMID 11232168
- [Background] Wiesner R, Rabkin J, Klintmalm G, McDiarmid S, Langnas A, Punch J, McMaster P, Kalayoglu M, Levy G, Freeman R, Bismuth H, Neuhaus P, Mamelok R, Wang W. A randomized double-blind comparative study of mycophenolate mofetil and azathioprine in combination with cyclosporine and corticosteroids in primary liver transplant recipients. Liver Transpl. 2001 May;7(5):442-50. doi: 10.1053/jlts.2001.23356. PMID 11349266
- [Background] Shaw LM, Korecka M, Venkataramanan R, Goldberg L, Bloom R, Brayman KL. Mycophenolic acid pharmacodynamics and pharmacokinetics provide a basis for rational monitoring strategies. Am J Transplant. 2003 May;3(5):534-42. doi: 10.1034/j.1600-6143.2003.00079.x. No abstract available. PMID 12752309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were current patients from 3 outpatient transplant offices and recruited between July 2006 and May 2008.
Pre-assignment Details: Participants were screened over a 2 week period. Three participants withdrew consent after signing the consent form. One participant failed screening (didn't attain threshold MPA level). These subjects were excluded from the trial before assignment to groups.
Groups:
- MMF, CNI Discontinued: Received Mycophenolate Mofetil (MMF); Complete withdrawal of calcineurin inhibitors (CNI)
- MMF; CNI Decreased: Received Mycophenolate Mofetil (MMF); calcineurin inhibitors (CNI) decreased to 50% of pre-enrollment dosage
Period: Overall Study
Arm/Group | MMF, CNI Discontinued | MMF; CNI Decreased
Started | 9 | 10
Completed | 6 | 9
Not Completed | 3 | 1
Not completed — Physician Decision | 2 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MMF, CNI Discontinued | MMF; CNI Decreased | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 10 | 17
  >=65 years | 2 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 56.11 (8.46) | 54.6 (7.26) | 55.32 (7.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 7 | 7 | 14
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Number of Biopsy Proven Rejections at 12 Months
Description: assessed by liver biopsy using Banff International Consensus Schema
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | MMF, CNI Discontinued | MMF; CNI Decreased
Number analyzed (Participants) | 6 | 9
participants | 0 | 0

2. Secondary Outcome: Patient and Graft Survival at 12 Months
Time Frame: 12 months
Population: everyone enrolled who completed the study
Measure: Number; unit: participants
Groups:
- CNI Discontinued: complete withdrawal of calcineurin inhibitors (CNI)
- CNI Reduction: calcineurin inhibitors (CNI) decreased to 50% of pre-enrollment
Arm/Group | CNI Discontinued | CNI Reduction
Number analyzed (Participants) | 6 | 9
participants | 6 | 9

3. Secondary Outcome: Number of Participants With Adverse Events Including Infections at 12 Months
Time Frame: 12 months
Population: everyone enrolled who completed the study
Measure: Number; unit: participants
Arm/Group | MMF, CNI Discontinued | MMF; CNI Decreased
Number analyzed (Participants) | 6 | 9
participants | 2 | 1

ADVERSE EVENTS:
Arm/Group | MMF, CNI Discontinued | MMF; CNI Decreased
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/10
Other Adverse Events (participants affected / at risk) | 9/9 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMF, CNI Discontinued (N=9) | MMF; CNI Decreased (N=10)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation alter with diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
change in white blood cell count (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MMF, CNI Discontinued (N=9) | MMF; CNI Decreased (N=10)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 6 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Increased liver enzymes (Hepatobiliary disorders) | 2 (3) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No